CLINICAL TRIAL: NCT01176838
Title: A Prospective Study on Newly Diagnosed Breast Cancer Patients: A 5 Year Follow Up on Quality of Life
Brief Title: A 5 Year Follow-up on Newly Diagnosed Breast Cancer Patients
Status: Terminated | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: IRB00007317
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-06

CONDITIONS: Newly Diagnosed Breast Cancer
Keywords: Breast Cancer Quality of Life Survey

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to provide the physicians with quality long term follow up data on subjects from the Breast Cancer Clinic and the Plastic Surgery Clinic who have been newly diagnosed with breast cancer and will receive treatment for the cancer at this facility. Over the last two decades many studies have been done concerning the quality of life after a mastectomy and/or reconstruction process. The majority of these studies only run for one year post reconstruction, some however, do include a two year follow up. The investigators are proposing a 5 year long term follow up study on subjects who will be diagnosed and treated here at the Breast Cancer Clinic and the Plastic Surgery Clinic. The investigators first questionnaire will be given prior to any treatment for breast cancer, giving us a baseline for the subject's current quality of life. At each successive year, the subject will be given another questionnaire with regards to their progression through the reconstructive process. At the end of 5 years, the subject will complete a final questionnaire. These questionnaires will deal with many areas of daily life functions; activities of daily living, anxiety, depression, social interactions, personal and sexual relationships.

DETAILED DESCRIPTION:
Upon informed consent of subject, a baseline questionnaire will be completed by the subject. At years 1, 2, 3, and 4 follow up questionnaires will be sent for completion to the subject. At year 5 a final questionnaire will be sent to the subject for completion.After all subjects have completed the study, data will be sent to the Department of Biostatics for analysis.

ELIGIBILITY:
Inclusion Criteria:

Any female age 18 or over that has been diagnosed with breast cancer and has been treated and followed in the Breast Cancer Clinic and the Plastic Surgery Clinic is eligible for study participation.

Exclusion Criteria:

Any person not meeting these requirements will not be eligible for study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of females ages 18 and over that have been newly diagnosed with breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R David, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Department of Plastic & Reconstructive Surgery, Winston-Salem, North Carolina, United States